CLINICAL TRIAL: NCT02768350
Title: Efficacy and Ventilatory Responsiveness of Ventilator Hyperinflation Technique to Re-expand Lung Atelectasis and Improved Airway Clearance on Patients With Critical Trauma Who Are Intubated and Mechanically Ventilated
Brief Title: Efficacy and Ventilatory Responses to VHI in Atelectasis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Guntaragorn Hongrattana, school of physical therapy, faculty of associated medical sciences, Khon Kaen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VHI-efficacy-atelectasis
Record Dates: First submitted 2016-02-02; First posted 2016-05-11 (Estimated); Last update posted 2018-03-09 (Actual); Status verified 2018-03

CONDITIONS: Atelectasis
Keywords: lung collapse; ventilator hyper inflation; hemodynamic responses; ventilatory responses; trauma patients
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group (Experimental): All of the participants in control group will be treated with conventional treatment for 3 days, The conventional treatments consist of: (1) Passive chest mobilization, (2) Positioning, (3) Side lying (good lung down), (4) Vibration. The conventional treatment consists of three consecutive periods; (1) baseline period: 10 minutes, (2) intervention period, and (3) recovery period: 10 minutes.
  Interventions: Procedure: Conventional treatment
- Experimental group (Experimental): All of the participants of the experimental group will be treated with ventilator hyperinflation technique (VHI) for 3 days. Tidal volume will increase from baseline (100% VT) to the tidal volume target at 1.5 times (150% VT). At this level, patients will receive six breathes and in each breathe will be sustained for 5 second (6 hyperinflation breathe per set); expiratory VT will return to baseline after each breath. Four sets of hyperinflation breathing will be used. After this, VT will decrease to baseline and patients have a 60 second for rest between hyperinflation set. The ventilator hyperinflation technique (VHI) consists of three consecutive periods; (1) baseline period: 10 minutes, (2) intervention period, and (3) recovery period: 10 minutes.
  Interventions: Procedure: Ventilator hyperinflation technique

INTERVENTIONS:
Procedure: Ventilator hyperinflation technique — Hyperinflation using a ventilator or "ventilator hyperinflation technique (VHI)" was developed from the manual hyperinflation (MHI) technique. There is no need to disconnect the patient when using the VHI technique and consequently there is no loss of PEEP and little or no risk of the adverse effects associated with MHI.
  Arms: Experimental group
Procedure: Conventional treatment — Conventional treatments are the routine treatment that patients were received from the physical therapist who take care them. The routine treatments are consist of chest physical therapy techniques (i.e. vibration, positioning, etc.) and others treatment (i.e. passive movement).
  Arms: Control group

SUMMARY:
The purpose of this study include (1) To investigate the efficacy of ventilator hyperinflation technique to re-expand lung atelectasis on patients with critical trauma who intubated and mechanical ventilation in the intensive care unit, (2) To investigate the effectiveness of ventilator hyperinflation technique to improve airway clearance on patients with critical trauma in the intensive care unit, and (3) To explore the acute responses of ventilatory functions to ventilator hyperinflation technique on patients with critical trauma who intubated and mechanical ventilation in the intensive care unit.

ELIGIBILITY:
Inclusion Criteria:

* Critical trauma patients with pulmonary complications who were intubated and mechanical ventilation and have a diagnosis of lobar atelectasis and/or plate-like atelectasis (atelectasis demonstrated on chest X-ray) will be considered for inclusion. For the sign of plate-like atelectasis will be persist on chest X-ray for 2 day
* The injuries may occur alone or combination of these injuries: 1) head injury, 2) chest injuries, including broken ribs, with or without hemothorax, pneumothorax and hemopneumothorax with intercostal chest drainage (ICD), 3) blunt abdominal, and 4) fracture of the limbs and/or spine.

Exclusion Criteria:

* acute respiratory distress syndrome (ARDS)
* acute lung injury (ALI)
* pulmonary contusion
* undrained pneumothorax, hemothorax, and hemopneumothorax
* bronchospasm
* pulmonary bullae/blebs
* lung tumors
* lung abscess
* haemoptysis
* mean arterial pressure (MAP) <70 mmHg
* positive end expiratory pressure (PEEP) >6 cmH2O
* heart rate (HR) >140 beats/min
* blood pressure (BP) <90/60 or >180/100 mmHg
* restlessness
* oxygen saturation (SpO2) <90%
* spontaneous respiratory rate (RR) >35 beats/min

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2016-05; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Chest Radiography | "Change from Baseline in Chest Radiography at Day 1 after Received Intervention (VHI)" and "Change from Baseline in Chest Radiography at Day 3 after Received Intervention (VHI)"
  The study took three day, chest radiography will be taken at 2 day before the study begin (first film; base line) and after day 1 (second film) and day 3 of the study (third film).
  Any improvement will be assessed by comparing the second and the third film to the first film by a radiologist who will be blinded to the treatment given.
  Atelectasis will grade using the following rating scale: 0 = no atelectasis; 1 = plate-like atelectasis; 2 = mild lobar collapse; 3 = moderate lobar collapse; and 4 = complete lower lobar collapse. Separate results will comply for the left and right lungs.

SECONDARY OUTCOMES:
Change from baseline in respiratory rate (RR) at during and end of ventilator hyperinflation technique (VHI) | Within 10 minutes before VHI, 8 minutes during VHI and 10 minute after VHI.
  Data will be recorded at 09.00, 09.02, 09.04, 09.06, 09.08, and 09.10 am for pre-intervention period, at 09.12, 09.14, 09.16, and 09.18 am for during intervention period (4 set of 6 VHI breath; each set take time about 2 min), and at 09.20, 09.24, 09.26, 09.28, and 09.30 am for post-intervention period.
  Data will be repeated record at the same time on day 2 and 3. Respiratory rate (RR) will be recorded from the display of mechanical ventilator.
Change from baseline in tidal volume (VT) at during and end of ventilator hyperinflation technique (VHI)hyperinflation technique (VHI) | Within 10 minutes before VHI, 8 minutes during VHI and 10 minute after VHI.
  Data will be recorded at 09.00, 09.02, 09.04, 09.06, 09.08, and 09.10 am for pre-intervention period, at 09.12, 09.14, 09.16, and 09.18 am for during intervention period (4 set of 6 VHI breath; each set take time about 2 min), and at 09.20, 09.24, 09.26, 09.28, and 09.30 am for post-intervention period.
  Data will be repeated record at the same time on day 2 and 3. Respiratory rate (RR) will be recorded from the display of mechanical ventilator.
Change from baseline in minute ventilation (VE) at during and end of ventilator hyperinflation technique (VHI)technique (VHI)hyperinflation technique (VHI) | Within 10 minutes before VHI, 8 minutes during VHI and 10 minute after VHI.
  Data will be recorded at 09.00, 09.02, 09.04, 09.06, 09.08, and 09.10 am for pre-intervention period, at 09.12, 09.14, 09.16, and 09.18 am for during intervention period (4 set of 6 VHI breath; each set take time about 2 min), and at 09.20, 09.24, 09.26, 09.28, and 09.30 am for post-intervention period.
  Data will be repeated record at the same time on day 2 and 3. Respiratory rate (RR) will be recorded from the display of mechanical ventilator.
Change from baseline in oxygen saturation (SpO2) at during and end of ventilator hyperinflation technique (VHI)hyperinflation technique (VHI)technique (VHI)hyperinflation technique (VHI) | Within 10 minutes before VHI, 8 minutes during VHI and 10 minute after VHI.
  Data will be recorded at 09.00, 09.02, 09.04, 09.06, 09.08, and 09.10 am for pre-intervention period, at 09.12, 09.14, 09.16, and 09.18 am for during intervention period (4 set of 6 VHI breath; each set take time about 2 min), and at 09.20, 09.24, 09.26, 09.28, and 09.30 am for post-intervention period.
  Data will be repeated record at the same time on day 2 and 3. Respiratory rate (RR) will be recorded from the display of mechanical ventilator.
Change from baseline in dynamic lung compliance (Cdyn) at during and end of ventilator hyperinflation technique (VHI) | Within 10 minutes before VHI, 8 minutes during VHI and 10 minute after VHI.
  Data will be recorded at 09.00, 09.02, 09.04, 09.06, 09.08, and 09.10 am for pre-intervention period, at 09.12, 09.14, 09.16, and 09.18 am for during intervention period (4 set of 6 VHI breath; each set take time about 2 min), and at 09.20, 09.24, 09.26, 09.28, and 09.30 am for post-intervention period.
  Data will be repeated record at the same time on day 2 and 3. Respiratory rate (RR) will be recorded from the display of mechanical ventilator.
Change from baseline in end-tidal pressure of carbon dioxide (PETCO2) at during and end of ventilator hyperinflation technique (VHI) | Within 10 minutes before VHI, 8 minutes during VHI and 10 minute after VHI.
  Data will be recorded at 09.00, 09.02, 09.04, 09.06, 09.08, and 09.10 am for pre-intervention period, at 09.12, 09.14, 09.16, and 09.18 am for during intervention period (4 set of 6 VHI breath; each set take time about 2 min), and at 09.20, 09.24, 09.26, 09.28, and 09.30 am for post-intervention period.
  Data will be repeated record at the same time on day 2 and 3. Respiratory rate (RR) will be recorded from the display of mechanical ventilator.
Change from baseline in peak inspiratory pressure (PIP) at during and end of ventilator hyperinflation technique (VHI) | Within 10 minutes before VHI, 8 minutes during VHI and 10 minute after VHI.
  Data will be recorded at 09.00, 09.02, 09.04, 09.06, 09.08, and 09.10 am for pre-intervention period, at 09.12, 09.14, 09.16, and 09.18 am for during intervention period (4 set of 6 VHI breath; each set take time about 2 min), and at 09.20, 09.24, 09.26, 09.28, and 09.30 am for post-intervention period.
  Data will be repeated record at the same time on day 2 and 3. Respiratory rate (RR) will be recorded from the display of mechanical ventilator.
Change from baseline in arterial blood gases (ABG) at end of ventilator hyperinflation technique (VHI) | Within one hour before VHI and 10 minute after VHI.
  Data will be recorded at 08.00 and 09.10 am for pre-intervention and post-intervention, respectively.
  Five milliliter of arterial blood will be collected from arterial line (A-line) for the analysis of arterial blood gases analysis (ABG).
24 hour sputum collection | The secretion will be collected 24 hours in each day.
  Endotracheal/tracheal suction will take at 08.30, 09.35, 11.00, 13.00, 15.00, 17.00, 19.00, 21.00, 23.00, 01.00, 03.00, 05.00, and 07.00 (24 hour). Sputum volume and wet weight at each time's collect will accumulate to represent for 24 hour sputum collection.
  The mucus secretion will be collected by nursing staff using sterile suctioning technique via tracheostomy (TT) or endotracheal (ET) tube, without adding any saline or sterile water.
Clearance index | Sputum content that collects at 08.30 and 09.35 will test by cough transportability method and compare between time point for represent the clearance index (at 08.30 for pre-intervention period and at 09.35 for post-intervention period).

CONTACTS AND LOCATIONS:
Locations (1):
- Khon Kaen University, Khon Kaen, Thailand